CLINICAL TRIAL: NCT02979496
Title: The Effect of Citrus Beverages on Gastrointestinal Function in Healthy Adults: a Randomized, Double-blind, Controlled Clinical Trial
Brief Title: Citrus Beverages and Gastrointestinal Function
Acronym: POM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: PepsiCo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB201602073
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: immune; citrus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0 g pomace (control) (Other): 16 oz of juice containing 0 g of citrus pomace will be consumed each day for 3 weeks by participants in the group receiving this assignment (group is unknown, double-blinded).
  Interventions: Dietary Supplement: 0 g pomace (control)
- 90 g pomace (Experimental): 16 oz of juice containing 90 g of citrus pomace will be consumed each day for 3 weeks by participants in the group receiving this assignment (group is unknown, double-blinded).
  Interventions: Dietary Supplement: 90 g pomace
- 180 g pomace (Experimental): 16 oz of juice containing 180 g of citrus pomace will be consumed each day for 3 weeks by participants in the group receiving this assignment (group is unknown, double-blinded).
  Interventions: Dietary Supplement: 180 g pomace
- Flavored water (control) (Other): 16 oz of a flavored, calorie-matched water beverage will be consumed each day for 3 weeks by participants in the group receiving this assignment (group is unknown, double-blinded).
  Interventions: Dietary Supplement: Flavored water (control)

INTERVENTIONS:
Dietary Supplement: 0 g pomace (control) — 16 oz of juice containing 0 g of citrus pomace will be consumed each day for 3 weeks by participants in the group receiving this assignment (group is unknown, double-blinded)
  Arms: 0 g pomace (control)
Dietary Supplement: 90 g pomace — 16 oz of juice containing 90 g of citrus pomace will be consumed each day for 3 weeks by participants in the group receiving this assignment (group is unknown, double-blinded).
  Arms: 90 g pomace
Dietary Supplement: 180 g pomace — 16 oz of juice containing 180 g of citrus pomace will be consumed each day for 3 weeks by participants in the group receiving this assignment (group is unknown, double-blinded).
  Arms: 180 g pomace
Dietary Supplement: Flavored water (control) — 16 oz of a flavored, calorie-matched water beverage will be consumed each day for 3 weeks by participants in the group receiving this assignment (group is unknown, double-blinded).
  Arms: Flavored water (control)

SUMMARY:
The purpose of this study is to evaluate the effect of daily intake of orange pomace on gastrointestinal function as measured by stool frequency. Additional outcomes will include aspects of digestive health, diet quality, and fasting blood glucose and lipid concentrations. Possible explanations for the mechanism of the pomace will be explored in microbial ecology analyses.

DETAILED DESCRIPTION:
In this randomized, double-blind, controlled trial, healthy adults will be asked to consume daily servings of orange juice containing either 0 g (n=120; control) or 180 g (i.e. 10 g fiber; n=120) of orange pomace for 3 weeks to assess the effect of the pomace on stool frequency. Blood samples will be obtained to assess the effect of the pomace on metabolic markers. Stool samples will be collected for analyses of the effect of the pomace on fecal bacteria known to be associated with health benefits (e.g., bifidobacteria). For exploratory analyses, additional groups will be asked to consume orange juice containing 90 g of pomace (i.e. 5 g fiber; n=40) or orange-flavored, calorie-matched water (n=40); outcomes from the water group will be compared to those of the 0 g pomace juice group to assess any effects of the juice alone, and outcomes from the 90 g pomace group will be compared to those of the 180 g and 0 g groups in microbiota analyses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-60 years of age
* Willing and able to consume 16 oz. of a citrus beverage daily for the 3-week study intervention
* Willing and able to avoid consumption of any orange, grapefruit, tomato or V-8 juice and whole oranges or grapefruits during the two weeks leading up to the study and during the study, not including the study beverage
* Willing and able to complete daily questionnaires online regarding dietary intake and general health and well-being, including gastrointestinal habits Note: we will recruit participants who will have Internet access for the duration of the protocol, but understand that, once enrolled, situations may change. If this is the case, paper copies of the online forms will be provided
* Willing to discontinue any prebiotic, probiotic, and fiber supplements after consenting
* Willing to provide blood via finger prick and a stool sample twice each, once at the beginning and once at the end of the study

Exclusion Criteria:

* Women who are lactating, know that they are pregnant, or are attempting to get pregnant
* Currently being treated for any physician-diagnosed diseases or conditions
* Vegetarians/vegans

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 330 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2017-04-29 (Actual); Study Completion 2017-04-29 (Actual)

PRIMARY OUTCOMES:
Change in Stool Frequency | Weeks -1,0,1,2,3
  The average number of stools per week compared between intervention groups.

SECONDARY OUTCOMES:
Change in Stool frequency as a function of stool consistency | Change from Weeks -1,0,1,2,3
  The average number of stools per week compared between intervention groups, including Bristol Stool Score category (stool types 1-7 with 1 = hard and 7 = liquid ) as a covariate in the statistical model.
Change in Diarrhea symptom score | Change from Weeks -1,0,1,2,3
  Measured By Gastrointestinal Symptom Response Scale (GSRS). Questionnaire asks participants about the previous seven days. Scores range from 1 (no discomfort) to 7 (very severe discomfort); lower scores are more desirable.
Change in Constipation symptom score | Change from Weeks -1,0,1,2,3
  Measured By Gastrointestinal Symptom Response Scale (GSRS). Questionnaire asks participants about the previous seven days. Scores range from 1 (no discomfort) to 7 (very severe discomfort); lower scores are more desirable.
Change in Indigestion symptom score | Change from Weeks -1,0,1,2,3
  Measured By Gastrointestinal Symptom Response Scale (GSRS). Questionnaire asks participants about the previous seven days. Scores range from 1 (no discomfort) to 7 (very severe discomfort); lower scores are more desirable.
Change in Reflux symptom score | Change from Weeks -1,0,1,2,3
  Measured By Gastrointestinal Symptom Response Scale (GSRS). Questionnaire asks participants about the previous seven days. Scores range from 1 (no discomfort) to 7 (very severe discomfort); lower scores are more desirable.
Change in Abdominal pain symptom score | Change from Weeks -1,0,1,2,3
  Measured By Gastrointestinal Symptom Response Scale (GSRS). Questionnaire asks participants about the previous seven days. Scores range from 1 (no discomfort) to 7 (very severe discomfort); lower scores are more desirable.
Change in Number of bifidobacteria in fecal samples | Change from Weeks 0 and 3
  Bifidobacteria in fecal samples will be quantified via quantitative polymerase chain reaction (qPCR) and compared between groups.
Change in Fasting blood glucose | Change from Weeks 0 and 3
  Fasting blood glucose determined by Cholestech assay

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, RD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No